CLINICAL TRIAL: NCT04621214
Title: Innovation of Audio-Visual Triage System in Combating the Spread of COVID-19 Infection and Its Efficacy: A Novel Strategy
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Dr Muhammad Mansoor Hafeez, Assistant Professor, University of Lahore
Other Study IDs: IRBEC/BIH/013-2020
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Audio-Visual Triage System; Anxiety Levels; COVID-19 Spread; GAD-7 Score; Healthcare Professionals; Screening Strategy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-A: Group A were performing their duties on visual triage
  Interventions: Device: Audio-Visual Triage System (AVT)
- Group-B: Group A were performing their duties on Audio-visual triage
  Interventions: Device: Audio-Visual Triage System (AVT)

INTERVENTIONS:
Device: Audio-Visual Triage System (AVT) — Audio System was added to visual triage that resulted in an AVT. Protocols of AVT included, a medical personal sits on TRIAGE DESK (with glass barrier sheet on it) wearing personal protective equipment (PPE) at a distance of more than 6 feet from the PATIENT DESK. Both desks are connected with Non-touchable MIC SYSTEM for communication

SUMMARY:
During the novel coronavirus pandemic, also known as SARS-CoV-2 or COVID-19 pandemic, frontline healthcare professionals suffered psychological as well as pathological trauma due to the lack of preparation to cope with this unforeseen situation. The protocols to prevent the spread of this disease proved to be less effective than anticipated. In these circumstances, improvement of the existing triage system was felt and an AUDIO-VISUAL TRIAGE (AVT) system was introduced to enhance confidence as well as increase the safety of frontline healthcare professionals. The current analysis was performed from March 21, 2020, to April 28, 2020, until the completion of sixty response forms, at Bahria Town International Hospital, Lahore. Thirty participants (Group A) deployed on visual triage and other thirty (Group B) on Audio-Visual triage for screening suspected cases of COVID-19 infection. Anxiety levels were measured by using the GAD-7 scoring system and the participants of both groups were periodically tested for COVID-19 infection by PCR. Independent t-test was used to evaluate the significance of different variables at a confidence level of 95%.

DETAILED DESCRIPTION:
A novel strategy 'Audio-Visual Triage' was introduced to boost up the confidence levels, lower down the anxiety levels and the most important factor is to reduce the risk of COVID-19 infection spread. This Triage system included Audio system to communicate with patients and access the COVID-19 infection status at recommended distance of 6 feet. The main disturbing factors that were noted on Visual triage system were, 1). Close contact of healthcare professionals with patients and attends, 2). Fear of transmission of infection lead to higher levels of anxiety. To assess the efficiency of AVT Anxiety level were analyzed by using Spitzer et al., 2006, General Anxiety Disorder-7 (GAD-7) scoring system and outcomes were assessed where a score less than 5 is taken as no anxiety, 5-9 interpreted as mild anxiety, 10-14 moderate anxiety, and ≥ 15 as severe anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Participants performing their duty on visual triage.

Exclusion Criteria:

* Those participants having previous psychological illness, frequently used to use the washroom, had non-serious attitude and poor compliance with the protocols of wearing PPEs were excluded from the study.

Ages: 20 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asymptomatic Healthy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Polymerase chain reaction (PCR) to detect SARS-CoV-2 virus | 12-24 hours
  Every participant was test for COVID-19 infection by PCR. At the end of the study we compare the Number of participant infected by Corona virus in Both groups.
General Anxiety Disorder-7 (GAD-7) scoring system | 15 - 20 minutes
  The GAD-7 is used to measure the severity of anxiety. Score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
  Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD. It is moderately good at screening three other common anxiety disorders - panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%) and post-traumatic stress disorder (sensitivity 66%, specificity 81%

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No